CLINICAL TRIAL: NCT06848881
Title: Cryoablation Versus Thoracoscopic Surgery for Pulmonary Ground-Glass Nodules: A Prospective, Randomized Controlled Trial
Brief Title: Cryoablation vs Thoracoscopic Surgery for GGN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director, Department of Respiratory Endoscopy, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHCHE202501
Record Dates: First submitted 2025-02-07; First posted 2025-02-27 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Ground-Glass Opacity
MeSH Terms: interventions — Cryosurgery; Thoracoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryoablation group (Experimental): Ground-glass nodules were treated using cryoprobe by bronchoscope.
  Interventions: Procedure: Cryoablation
- Thoracoscopic Surgery group (Active Comparator): Ground-glass nodules were treated by video-assisted thoracoscopic surgery (VATS). Based on the location of the GGN, select the appropriate surgical resection range (wedge resection, segmentectomy, lobectomy, or combined segmentectomy).
  Interventions: Procedure: Thoracoscopic Surgery

INTERVENTIONS:
Procedure: Cryoablation — The eligible patient will be randomized to cryoablation group to receive cryoablation.
  Arms: Cryoablation group
Procedure: Thoracoscopic Surgery — The eligible patient will be randomized to thoracoscopic surgery group to receive surgery.
  Arms: Thoracoscopic Surgery group

SUMMARY:
The aim of this study is to investigate the efficacy and safety of Cryoablation and Thoracoscopic Surgery in the treatment of pulmonary ground-glass nodules.

DETAILED DESCRIPTION:
The primary treatment for GGN type lung cancer is surgical resection, typically using video-assisted thoracoscopic surgery (VATS). Image-guided ablation therapy is considered as a treatment option for early-stage lung cancer patients unsuitable for surgery. It has been recommended by several guidelines as one of the curative treatment methods for primary lung cancer. Among various ablation techniques, cryoablation has the lowest complication rate. However, there is currently no research exploring whether cryoablation is not inferior to thoracoscopic surgery in terms of safety and efficacy in treating highly suspected malignant lung GGNs. This study was designed as a prospective, randomized controlled trial, with 160 patients expected to be enrolled in the study, randomized in a 1:1 ratio to cryoablation and thoracoscopic surgery treatment groups. The primary endpoint is the 2-year disease-free survival. Secondary endpoints include 1-month mortality rate, overall survival, 5-year disease-free survival, local recurrence rate, VATS/ cryoablation completion rate, safety, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years old.
2. The size of the GGN was 6-20mm (with less than 25% solid component), and the number of nodules requiring treatment in the short term is less than 3.
3. Pathological confirmation of the GGN as non-small cell lung cancer; or progression of the GGN during at least 3 months of follow-up, including enlargement of the largest diameter, increase in solid component, or the appearance of a significant solid component in a previously pure GGN, with multidisciplinary discussion (including radiology, thoracic surgery, and pulmonology) suggesting malignancy.
4. No lymph node, pulmonary, or distant metastasis to other organs.
5. After multidisciplinary evaluation, the patient is considered capable of tolerating both surgical and ablation procedures.
6. Unsuitable for radiation therapy or refuses radiation therapy.
7. Willing to participate in this clinical study and sign the informed consent form.

Exclusion Criteria:

1. Patients in poor general condition, with ECOG physical fitness score >2, unable to tolerate surgery or ablation therapy, or with relevant contraindications.
2. Patients who have previously received other treatments for pulmonary GGNs.
3. Patients with poor compliance.
4. Severe heart, lung, kidney, brain, or other vital organ diseases.
5. Active bacterial or fungal infections.
6. Simultaneous or metachronous (within the past 5 years) double cancers.
7. Women during pregnancy or breast-feeding.
8. History of prior lung surgery or radiation therapy.
9. Bleeding tendency, abnormal coagulation functions, or coagulation disorders that cannot be corrected after treatment.
10. Contraindications to general anesthesia.
11. Expected survival time < 6 months.
12. The researcher believes that it is not suitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2030-04-15 (Estimated); Study Completion 2030-04-15 (Estimated)

PRIMARY OUTCOMES:
2-year disease-free survival | Up to 2 years
  Defined as the time from enrollment to the occurrence of disease recurrence, the discovery of new lesions, or death due to any cause.

SECONDARY OUTCOMES:
1-month mortality rate | 1 month after the treatment
  The proportion of patients who die within one month after treatment.
Overall survival | Up to 2 years, 5years
  Defined as the time from enrollment to death from any cause, or to the last contact with surviving patients.
5-year disease-free survival | Up to 5 years
  Defined as the time from enrollment to the occurrence of disease recurrence, the discovery of new lesions, or death due to any cause.
Local recurrence rate | Up to 5 years
  The proportion of patients who experience disease recurrence at the original treatment site.
VATS/ cryoablation completion rate | immediately after the treatment
  The proportion of patients in whom VATS or cryoablation is successfully completed.
Forced Expiratory Volume in 1 Second (FEV1) | 3 months after the treatment
  The maximum volume of air exhaled in the first second during a forced expiration following maximal inhalation.
Forced Vital Capacity (FVC) | 3 months after the treatment
  The total volume of air exhaled as forcefully and completely as possible after maximal inhalation.
Adverse events and serious adverse events | 3 months after the treatment
  Complications at 3 months after the treatment will be assessed using the Clavien-Dindo classification of surgical complications.
  Aderse events will be evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Quality of life assessment | 1 week after the treatment
  Pain scores.
Length of hospital stay | 1 month after the treatment
  The duration of hospital stay after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, MD, PhD, Study Director — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No